CLINICAL TRIAL: NCT06512350
Title: Using Infrared Spectroscopy to Analyze Volatile Organic Compounds in the Breath of Patients With Breast Cancer
Brief Title: Identifying Patterns in the Breath of Individuals With Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Breathe BioMedical Inc (Industry)
Collaborators: Mayo Clinic (Other); George Washington University (Other); Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: BBMCP2024
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Dense Breast Tissue; Infrared Spectroscopy; Machine Learning
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Breast Cancer Cohort: Subjects with mammography-confirmed dense breast tissue (BI-RADS density score of C or D) and with biopsy-proven primary breast cancer.
- Control Cohort: Subjects with mammography-confirmed dense breast tissue (BI-RADS density score of C or D) and a negative MRI (for surveillance or diagnostic purposes with BI-RADS 1 or 2) that confirms the absence of breast cancer.
- Breast Cancer Cohort - Surgery: Subjects with mammography-confirmed dense breast tissue (BI-RADS density score of C or D) and with biopsy-proven primary breast cancer, who have undergone surgery at Mayo Clinic Florida will be screened to provide a second breath sample. The second breath sample will be collected at least six months following the completion of all standard of care treatment (excluding adjuvant endocrine therapy and adjuvant HER2 directed monoclonal antibody such as trastuzumab).

SUMMARY:
Researchers will compare the breath profiles of women with breast cancer and those without to determine whether there are disease-specific patterns that can be leveraged to facilitate breast cancer detection.

Women with mammogram-confirmed dense breast tissues undergoing standard-of-care breast cancer screening will be invited to participate. Those who provide informed consent will provide one breath sample and fill out a questionnaire about their medical history with help from the research coordinators. Breath samples will be collected prior to standard of care biopsy or MRI, and patients will be stratified into the case or control group based on their test results.

The primary goal of this project is to use exhaled alveolar breath and the subsequent spectral data produced by Breathe BioMedical's cavity ring-down spectrometer to further develop Breathe BioMedical's technology and machine learning algorithms to determine the feasibility of detecting breast cancer in women with dense breast tissue.

Secondarily, this project aims to identify patterns of VOCs that are either over- or under-represented in participants with breast cancer when compared to the breath profiles of participants without breast cancer. This project will also assess performance characteristics of the technology (e.g. sensitivity, specificity, false negative rate, and false positive rate) including subgroup analyses. This project aims to understand intra-subject variability by exploring differences in breath signatures before and after definitive management of breast cancer, including surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* Female (sex as assigned at birth);
* Aged 40 - 74 years;
* Mammography confirmed dense breast tissue (BI-RADS density score of C or D);
* Scheduled for standard of care biopsy or MRI;
* Fluent in language of consent (English, Spanish, or French);
* Ability to give informed consent;
* Able to provide a breath sample.

Exclusion Criteria:

* Mammography confirmed fatty breast tissue (BI-RADS A or B);
* Prior history of breast cancer;
* Previous surgical biopsy or surgical excision of breast cancer in the past six months;
* History of cancer (except basal cell or squamous cell carcinoma of the skin) in the past year;
* Acute respiratory infection and/or symptoms in the past seven days;
* MRI BI-RADS 3 undergoing active surveillance (MRI requiring six-month follow-up).
* Pregnant or become pregnant during the study.

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population will be women aged 40-74 with dense breast tissue. Women who are scheduled for standard of care breast biopsy or MRI will be recruited, and breath will be collected prior to breast biopsy or MRI. Those with biopsy-proven primary breast cancer will be assigned to the case cohort (true positives). Subjects in this cohort who are proceeding to breast surgery at Mayo Clinic Florida will be screened to provide a second breath sample, 6 months after the completion of treatment. To be eligible for the control cohort, subjects must have a negative MRI (for surveillance or diagnostic purposes with BI-RADS 1 or 2) that confirms the absence of breast cancer (true negatives). Individuals who have received an MRI up to 8 weeks prior to breath sample collection may be approached, granted inclusion and exclusion criteria are met. Subjects will be recruited from participating clinical centers in Canada and the United States.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Compare the breath spectra from patients with breast cancer and from healthy controls using mathematical/statistical models to further develop Breathe BioMedical's technology and machine learning algorithms. | 12 months
  Using exhaled alveolar breath and the subsequent spectral data produced by Breathe BioMedical's infrared cavity ring-down spectrometer, the goal is to identify patterns of VOCs that are either over- or under-represented in the breath profiles of subjects with breast cancer compared to the breath profiles of healthy controls. Machine learning performance characteristics will also be assessed (e.g., sensitivity, specificity, false negative rate, and false positive rate) including subgroup analyses. This will allow for the determination of the feasibility of detecting breast cancer in women with dense breast tissue.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - GW Comprehensive Breast Center, Washington D.C., District of Columbia
  - Mayo Clinic Breast Clinic, Jacksonville, Florida
  - Duke University Medical Cente, Durham, North Carolina